CLINICAL TRIAL: NCT03229460
Title: High Flow Nasal Oxygen Therapy in Perioperative Period of the Adult With Hypercapnic and Hypoxemic Respiratory Faliure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Bin He, M.D./Ph.D., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-17-008
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Acute Respiratory Failure With Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- standard low flow therapy (Active Comparator): In the standard low flow therapy is applied continuously through a nonrebreather face mask at a flow rate of 10 liters per minute or more. The rate was adjusted to maintain an oxygen saturation level of 92% or more.
  Interventions: Other: standard low flow therapy
- high flow nasal oxygen therapy (Experimental): In the high-flow-oxygen group is passed through a heated humidifier and applied continuously through large-bore binasal prongs, with a gas flow rate of 30-60 liters per minute . The fraction of oxygen in the gas flowing in the system was subsequently adjusted to maintain an Spo2 of 92% or more.
  Interventions: Device: high flow nasal oxygen therapy
- Noninvasive ventilation (Placebo Comparator): In the noninvasive-ventilation group is delivered to the patient through a face mask that was connected to an ICU ventilator,with pressure support applied in a noninvasive ventilation mode. The Fio2 or PEEP level (or both) were then adjusted to maintain an Spo2 of 92% or more.
  Interventions: Device: association of high flow nasal oxygen therapy and non invasive positive pressure ventilation

INTERVENTIONS:
Other: standard low flow therapy — In the standard low flow therapy oxygen group, oxygen at a flow rate of 10 liters per minute or more.
  Arms: standard low flow therapy
Device: high flow nasal oxygen therapy — The patient will receive high flow nasal of humidified oxygen, set between 30 to 60 l/min. The inspired fraction of oxygen (FiO2) will be adjusted in order to obtain a SpO2 >92%.
  Arms: high flow nasal oxygen therapy
Device: association of high flow nasal oxygen therapy and non invasive positive pressure ventilation — The patient will receive successively in a day NPPV and O2-HFN. The NPPV will be applied with an airway humidification achieved by using a heated humidifier and a facial mask adapted to the morphology of the patient. The settings will be adjusted as follow : an inspiratory pressure between 6 to 14 cmH2O, in order to obtain a tidal volume between 7 to 10 ml/kg of predicted weight, a positive expiratory pressure between 0 to 10 cmH2O in order to obtain a SpO2 >92% with the minimal FiO2.
  Arms: Noninvasive ventilation

SUMMARY:
The purpose of this study is to determine the impact of hign-flow nasal therapy on the adult with hypercapnia and hpoxemia respiratory faliure in comparison with standard oxygen therapy ang noninvasive ventilation.

DETAILED DESCRIPTION:
Humidified high flow nasal oxygen therapy decreases dilution of the inhaled oxygen and, by matching patient's peak flow, allows accurate delivery of the set FiO2 throughout the whole inspiratory phase.The purpose of this study is to determine the impact of hign-flow nasal therapy on adult hypercapnic respiratory failure by comparing with nasal continuous positive airway pressure

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic and no hypercapnic acute respiratory failure :
* severe dyspnea at rest with a respiratory rate >25 breaths/min
* PaO2/FiO2 <300
* PaCO2 <45 mmHg,

Exclusion Criteria:

* age <18 years
* NPPV contraindications
* past history of respiratory chronic disease (COPD, cystic fibrosis…)
* cardiac pulmonary edema
* Pre-defined intubation
* other than respiratory organ failure : systolic pressure <90 mmHg,current treatment with epinephrine or norepinephrine, decreased level of consciousness ( Glasgow score ≤ 12)
* profound aplasia (white cells count <1000/mm 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the number of patients in each group who require endotracheal intubation with mechanical ventilation | 28days
  To compare the number of patients in each group who require endotracheal intubation with mechanical ventilation

SECONDARY OUTCOMES:
mechanical ventilation-free to day 28 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided